CLINICAL TRIAL: NCT05248295
Title: Investigating the Effects of Rhythm and Entrainment on Fluency in People With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Lauryn Zipse, Ph.D., CCC-SLP, Associate Professor, MGH Institute of Health Professions
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018P001160; R15DC019231 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-02-21 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Aphasia; Apraxia of Speech
MeSH Terms: conditions — Aphasia; Apraxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with aphasia (Experimental): Adults with stroke-based aphasia. Designating this group as experimental reflects the focus on studying responses in people with aphasia. All participants will complete the same 4 study conditions in a 2x2 design (Unison vs. Solo and Metrical vs. Conversational).
  Interventions: Behavioral: Unison speech (vs. solo); Behavioral: Metrical timing (vs. conversational)
- Healthy controls (Other): Adults without a history of speech, language, or neurological disorder, or stroke. This group is intended to serve as a context-providing reference group rather than a true comparator. All participants will complete the same 4 study conditions in a 2x2 design (Unison vs. Solo and Metrical vs. Conversational).
  Interventions: Behavioral: Unison speech (vs. solo); Behavioral: Metrical timing (vs. conversational)

INTERVENTIONS:
Behavioral: Unison speech (vs. solo) — Participants will repeat sentences in four conditions, in a 2x2 design with the factors unison vs. solo repetition, and metrical vs. conversational speech timing. Measures of speech accuracy and timing will be collected.
Behavioral: Metrical timing (vs. conversational) — This is the secondary contrast in the 2x2 design described above.

SUMMARY:
Speaking in unison with another person is included as a part of many treatment approaches for aphasia. It is not well understood why and how this technique works. One goal of this study is to determine who benefits from speaking in unison, and what characteristics of speech are most helpful. Another goal is to investigate a possible mechanism for this benefit: why does speaking in unison help? A possible mechanism for this benefit is examined, by testing whether the degree of alignment of a person's speech with that of another speaker can account for unison benefit.

DETAILED DESCRIPTION:
Aphasia is an acquired language disorder, most commonly due to stroke. It can affect an individual's ability to speak, understand spoken language, read, and write. Many treatments designed to improve spoken language in persons with aphasia (PWAs) use unison speech, having the person with aphasia speak along with the clinician or with a recording. One goal of this study is to determine who benefits from speaking in unison, and what characteristics of speech help them the most. Another goal is to investigate a possible mechanism for this benefit: why does speaking in unison help? This knowledge is important because understanding who benefits from this commonly used and potentially powerful therapy component, under which conditions they benefit, and why they do, is critical for customizing therapy so it can be as effective and efficient as possible. Unison speech is conducted using one of two different timing patterns: (1) a natural conversational pattern, which is used in everyday conversations, or (2) a metrical pattern, which follows a beat-based timing framework, as in songs or some poems. In either case, precisely aligning one's speech with that of another person (i.e., entraining one's speech) requires prediction: each speaker must plan their own speech motor commands before having heard the other speaker say the words they are planning. Natural conversational timing requires the speaker to make use of knowledge about language, particularly grammar, to align with the other person. In contrast, a metrical pattern allows a speaker to predict speech timing without relying heavily on language-based knowledge. Given that many PWAs have impaired grammar, we hypothesize that most PWAs will benefit more from speaking in unison to sentences with metrical vs. conversational timing patterns. However, there is great variation in linguistic, motor speech, and timing skills across PWAs, so metrical and conversational timing patterns are likely to have different degrees of effectiveness for different individuals. Results from this study will demonstrate how individual characteristics and speech timing affect whether or not a person with aphasia benefits from speaking in unison. Results will also indicate whether a speaker's ability to predict speech timing is necessary for a benefit of unison speech. Prediction ability will be measured by how closely the speaker aligns their speech with a spoken model.

ELIGIBILITY:
Inclusion Criteria:

* Native-speaker fluency in American English (prior to stroke for people with aphasia)
* Controls must report no history of speech, language, neurological disorders, or stroke
* People with aphasia must be at least 6-months post-stroke, and aphasia must be due to stroke

Exclusion Criteria:

* Inadequate hearing ability to reliably complete task: fail hearing screen
* Inadequate cognitive ability to understand and remember task: fail cognition screening (different measures for controls and people with aphasia)
* Inadequate speech repetition ability to complete task, or to be considered a control: fail speech repetition screening (different thresholds for controls and people with aphasia)
* Inadequate auditory comprehension ability to understand task: fail auditory comprehension screen (people with aphasia only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauryn Zipse, PhD, Principal Investigator — MGH IHP
Locations (1):
- MGH IHP, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- People With Aphasia: Adults with stroke-based aphasia
- Controls: Adults without a history of speech, language, or neurological disorder, or stroke
Period: Overall Study
Arm/Group | People With Aphasia | Controls
Started | 23 | 52
Completed | 18 | 49
Not Completed | 5 | 3
Not completed — found ineligible | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Data loss: audio recording error | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | People With Aphasia | Controls | Total
Number analyzed (Participants) | 23 | 52 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (7.6) | 42.4 (18.4) | 47.5 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 31 | 40
  Male | 14 | 21 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, not Hispanic | 20 | 36 | 56
  White, Hispanic | 0 | 1 | 1
  White, unknown ethnicity | 0 | 2 | 2
  Black, not Hispanic | 3 | 5 | 8
  Black, Hispanic | 0 | 0 | 0
  Black, unknown ethnicity | 0 | 0 | 0
  Asian, not Hispanic | 0 | 6 | 6
  Asian, Hispanic | 0 | 1 | 1
  Asian, ethnicity unknown | 0 | 0 | 0
  race not specified, ethnicity unknown | 0 | 1 | 1
Hearing Screen [Count of Participants; unit: Participants] — passed a hearing screening, demonstrating thresholds < 40 dB at 1 kHz, 2 kHz, and 4 kHz in at least one ear, tested in a quiet room
  Participants | 22 | 52 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percent Syllables Correct
Description: The percentage of syllables correctly repeated from the target sentences will be computed for each contrast, Unison vs. Solo and Metrical vs. Conversational, capturing all 4 conditions in the 2x2 design (Unison Metrical, Unison Conversational, Solo Metrical, Solo Conversational). A protocol will be used to score syllables for correctness.
Time Frame: 1 day study visit
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Controls | People With Aphasia
Number analyzed (Participants) | 49 | 18
percentage
  Unison | 99.22 (1.08) | 64.26 (23.13)
  Solo | 99.46 (1.18) | 52.71 (33.57)
  Metrical | 99.65 (0.67) | 60.47 (29.68)
  Conversational | 99.03 (1.39) | 56.50 (28.98)
Statistical Analysis 1: Comparison: People With Aphasia; People with aphasia (PWA) were not directly compared to controls since the finding of a lower % syllables correct in any condition in PWA would be trivial. Instead, within-groups analyses were conducted to understand how the experimental variables affected syllable accuracy within each group; Test type: Other — Separate regression models were used within each group (People with aphasia and Controls) to independently assess the effects of the variables. Below, the results are reported for the effect of production condition (Unison vs. Solo) for the group of interest, People with aphasia; p = 0.077, Regression, Logistic — Results are reported for production condition for people with aphasia (experimental group); Odds Ratio (OR) = 1.21, Standard Error of Mean 0.13 — OR computed with Unison as the numerator and Solo as the denominator
Statistical Analysis 2: Comparison: People With Aphasia; Test type: Other — Below, the results are reported for the effect of timing condition (Metrical vs. Conversational) for the group of interest, People with aphasia; p > .1, Regression, Logistic — Results are reported for Timing Condition for the People with aphasia
Statistical Analysis 3: Comparison: People With Aphasia; Test type: Other — Below, the results are reported for the interaction effect between production condition and timing condition for the group of interest, People with aphasia; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.55, Standard Error of Mean 0.13 — OR computed as ((Unison Metrical)/(Unison Conversational)) / ((Solo Metrical)/(Solo Conversational))
Statistical Analysis 4: Comparison: Controls; Separate regression models were used within each group. Here, the results are reported for the Control group; Test type: Other; p = 0.036, Regression, Logistic — Results are reported for Production Condition for the Control group; Odds Ratio (OR) = 0.63, Standard Error of Mean 0.14 — OR computed with Unison as the numerator and Solo as the denominator
Statistical Analysis 5: Comparison: Controls; Test type: Other — Below, the results are reported for the effect of timing condition (Metrical vs. Conversational) for the control group; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.36, Standard Error of Mean 1.19 — OR computed with Metrical as the numerator and Conversational as the denominator
Statistical Analysis 6: Comparison: Controls; Test type: Other — Below, the results are reported for the interaction effect between production condition and timing condition for the control group; p > .1, Regression, Logistic

2. Secondary Outcome: Mean Syllable Offset From Model
Description: Of the syllables attempted by the participant, the mean offset from the corresponding target syllable in the model is computed for each syllable for each participant using the formula (p - d) - s, where p is the timing of voicing onset in the participant response, d is the timing of voicing onset in the model, and s is the line delay in the audio equipment. Means are computed for each participant and each condition.
  Note this measure can only be computed in the Unison conditions (Unison Metrical and Unison Conversational), since the Solo conditions do not have a simultaneous spoken model to which the participant is trying to align their speech.
Time Frame: 1 day study visit
Population: Acoustic data were inadequate for 1 participant with aphasia (could not be reliably labeled due to vocal quality, resulting in too few data points for analysis for this participant).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Controls | People With Aphasia
Number analyzed (Participants) | 49 | 17
seconds
  Metrical | -.016 (.028) | 0.030 (0.052)
  Conversational | 0.006 (0.040) | 0.154 (0.188)
Statistical Analysis 1: Comparison: People With Aphasia; People with aphasia were not directly compared to Controls since the Control group is a context-providing reference group rather than a true comparator. Instead, within-groups analyses were conducted to understand how the experimental variable affected timing alignment in each group; Test type: Other — Separate regression models were used within each group (People with aphasia and Controls) to independently assess the effects of Timing Condition. Production Condition is not included in the analysis since all timing data are from the unison production condition, by definition; p < 0.001, Regression, Linear — Results are reported for people with aphasia (experimental group); Slope = -0.14, Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Controls; People with aphasia were not directly compared to Controls since the Control group is a context-providing reference group and not a true comparator. Instead, within-groups analyses were conducted to understand how experimental variables affected timing alignment in each group; Test type: Other; p < 0.001, Regression, Linear — Results are reported for the Control group; Slope = -0.05, Standard Error of Mean 0.00

ADVERSE EVENTS:
Time Frame: One study visit for controls and two study visits for people with aphasia, typically 1 day to 2 weeks apart
Groups:
- Intervention: All participants will repeat sentences under four speech conditions, in a 2x2 design
  Unison speech (vs. solo): Participants will repeat sentences in four conditions, in a 2x2 design with the factors unison vs. solo repetition, and metrical vs. conversational speech timing. Measures of speech accuracy and timing will be collected.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT05248295/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT05248295/ICF_001.pdf